CLINICAL TRIAL: NCT04485520
Title: Efficacy of the Extract of Carica Papaya as an Inhibitor of Streptococcus Mutans in Students of the Faculty of Dentistry in the Year 2018
Brief Title: Efficacy of the Extract of Carica Papaya as an Inhibitor of Streptococcus Mutans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julieta María Méndez Romero (Other)
Responsible Party: Sponsor-Investigator, Julieta María Méndez Romero, Head of Writting and Publication Department, Regional Health Research Institute, Universidad Nacional de Caaguazu
Organization: Universidad Nacional de Caaguazu (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00140
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Streptococcus, Other Specified Group; Dental Plaque
Keywords: Saliva; dental plaque; streptococcus mutans
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carica Papaya extract (Experimental): Carica Papaya at 3%
  Interventions: Other: CARICA PAPAYA MOUTHWASH
- Chlorhexidine (Active Comparator): 0.12% chlorhexidine mouthwash formulation (commercially available)
  Interventions: Other: CHLORHEXIDINE MOUTHWASH

INTERVENTIONS:
Other: CARICA PAPAYA MOUTHWASH — Each application was 10 ml. applied for 1 minute, once a day for 8 days
  Arms: Carica Papaya extract
Other: CHLORHEXIDINE MOUTHWASH — Each application was 10 ml. applied for 1 minute, once a day for 8 days
  Arms: Chlorhexidine

SUMMARY:
Papaya has effects on oral pathogenic microorganisms, it also has anticoagulant quality, amebicidal action, antimicrobial, bacteriostatic and antifungal activity on different bacteria, especially on Streptococcus mutans, this can be exploited in the dental area. The objective of the study was to determine the efficacy of Carica Papaya peel extract (suckling) as an inhibitor of Streptococcus Mutans in students of the dental faculty of the National University of Caaguazú in 2018.

DETAILED DESCRIPTION:
Specific objectives

* To determine the inhibition of the extract of the peel of Carica Papaya (baby) at 3% on Streptococcus Mutans by age and sex grouping.
* To quantify the inhibition of the extract of the peel of Carica Papaya (baby) at 3% on the growth of Streptococcus Mutans before, at 10 minutes and 8 days of use in the experimental group.
* Quantify the inhibition of 0.12% Chlorhexidine Gluconate on the growth of Streptococcus Mutans before, after 10 minutes and 8 days of use in the control group.
* Compare the count of Colony Forming Units (CFU) between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants that signed the informed consent

Exclusion Criteria:

* allergic to carica papaya
* ongoing medical or dental treatment that could interfere with the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-10-21 (Actual); Study Completion 2017-10-21 (Actual)

PRIMARY OUTCOMES:
Number of Colony Forming units (Stage 1) | thorough study completion, an average of 24 hours
  Before Intervention
Number of Colony Forming units (Stage 2) | 10 minutes after mouthwash use
  After Intervention
Number of Colony Forming units (Stage 3) | 8 days after mouthwash use
  After Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Diego Céspedes, Principal Investigator — Facultad de Odontología, Universidad Nacional de Caaguazu; Ulises A Villasanti Torales, Study Director — Facultad de Odontologia, Universidad Nacional de Caaguazu
Locations (1):
- Facultad de Odontología Universidad Nacional de Caaguazú, Coronel Oviedo, International, Paraguay

IPD SHARING:
Plan to Share IPD: Yes
By email
Supporting Information: Study Protocol, SAP
Time Frame: From the time the protocol is available in clinical trials.gov and with no limit of time
Access Criteria: Researchers that want to know about the study and use the protocol

REFERENCES:
- [Background] Saliasi I, Llodra JC, Bravo M, Tramini P, Dussart C, Viennot S, Carrouel F. Effect of a Toothpaste/Mouthwash Containing Carica papaya Leaf Extract on Interdental Gingival Bleeding: A Randomized Controlled Trial. Int J Environ Res Public Health. 2018 Nov 27;15(12):2660. doi: 10.3390/ijerph15122660. PMID 30486374